CLINICAL TRIAL: NCT03566602
Title: Single-arm, Open-label, Multicenter Study to Evaluate the Safety and Performance of Dura Sealant Patch in Reducing CSF Leakage Following Elective Cranial Surgery
Brief Title: Evaluate the Safety and Performance of Dura Sealant Patch in Reducing CSF Leakage Following Elective Cranial Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polyganics BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIP-1
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2019-03

CONDITIONS: Cerebrospinal Fluid Leak
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dura Sealant Patch (Other): Application of Dura Sealant Patch after closure of the dura mater
  Interventions: Device: Dura Sealant Patch

INTERVENTIONS:
Device: Dura Sealant Patch — Adjunctive bioresorbable patch

SUMMARY:
The objective of the study is to clinically assess the safety and performance of the Dura Sealant Patch as a means of reducing intra- as well as post-operative CSF leakage in patients undergoing elective cranial intradural surgery with a dural closure procedure.

ELIGIBILITY:
Inclusion Criteria:

Preoperative Subjects who are able to provide a written informed consent prior to participating in the clinical investigation.

Subjects who are ≥ 18 years old. Subjects who are able to comply with the follow-up or other study requirements. Subjects who are planned for an elective intracranial intradural surgery in whom a dural incision of at least 2 cm in length is necessary, which will be closed.

Female subjects of child bearing potential must agree to use any form of contraception from the time of signing the informed consent form through 90 days post-surgery.

Intraoperative Surgical wound classification Class I/Clean. Minimally 5 mm of dural space surrounding dural opening.

Exclusion Criteria:

Preoperative Female subjects who are pregnant or breastfeeding. Subjects with an assumed impaired coagulation due to medication or otherwise. Subjects suspected of an infection requiring antibiotics. Subjects with any type of dural diseases in planned dural closure area. Subjects requiring re-opening of planned surgical area within 90 days after surgery.

Subjects requiring local radiotherapy in planned surgical area. Subjects with a known allergy to any of the components of the Dura Sealant Patch.

Subject who previously participated in this study or any investigational drug or device study within 30 days of screening.

Subjects with a presence of hydrocephalus. Intraoperative Subjects in whom elevation of PEEP or pCO2 has a potential detrimental effect. Subjects who will require a CSF or wound drain, electrodes or other devices passing the dural layer or extra to intracranial bypass surgery.

Primary closure of the dura mater with synthetic, non-autologous or autologous material other than galea.

A gap > 3 mm after primary closure of the dura mater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Incidence of wound infection confirmed by increase of CRP and positive cultures | up to 30 days after surgery
  wound infection confirmed by increase of CRP and positive cultures
Incidence of intra-operative CSF leakage after patch application at 15 cmH2O of Positive End Expiratory Pressure (PEEP) | intra-operative
  intra-operative CSF leakage
Incidence of percutaneous CSF leak confirmed by β-2 transferrin test | up to 30 days after surgery
  Percutaneous CSF leak confirmed by β-2 transferrin test

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (2):
  - Elisabeth TweeSteden Ziekenhuis, Tilburg
  - UMCU, Utrecht
- University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Van Doormaal T, Germans MR, Sie M, Brouwers B, Carlson A, Dankbaar JW, Fierstra J, Depauw P, Robe P, Regli L. Single-arm, open-label, multicentre first in human study to evaluate the safety and performance of dural sealant patch in reducing CSF leakage following elective cranial surgery: the ENCASE trial. BMJ Open. 2021 Jul 28;11(7):e049098. doi: 10.1136/bmjopen-2021-049098. PMID 34321304